CLINICAL TRIAL: NCT04857320
Title: A Physician-Initiated Randomised, Multiple-Dose, Single Period, Phase II Dose Ranging Study to Examine Transdermal Human Insulin In Adult Healthy Volunteer Patients
Brief Title: Transdermal Insulin Response In Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Transdermal Delivery Solutions Corp (Industry)
Collaborators: Langford Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LEV 101-D-022521
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pharmacodynamic Response to Small Doses of Insulin
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Intervention Model Description: Healthy Males, aged 20 to 60, Non-diabetic and Hemoglobin A1c test results of less than 6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Main Experimental (Experimental): Each subject will receive doses applied to the skin of 0.075 IUs / Kilogram Body Weight, 0.1 IUs/Kilogram Body Weight and 0.15 IUs /Kilogram Body Weight
  Interventions: Combination Product: Human insulin

INTERVENTIONS:
Combination Product: Human insulin — Human Insulin from recombinant source delivered in a solution capable of enabling transdermal delivery formulated at 100 IU/mL of delivery vehicle.

SUMMARY:
Bio-fermentation produced Human insulin is available without prescription in the U.S. This study is a physician-initiated trial of a formula enabling transdermal delivery of human insulin.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the amount of lowering serum glucose as a function of dose of a topically applied formulation of Human Insulin administered by syringe measurement to adult Healthy Volunteer subjects as compared to no treatment. A 5-day period of daily blood sugar monitoring by means of wearable Continuous Glucose Monitor and insulin dosing for 3 days then monitoring for at least 3 days following will form the baseline and experimental data for each subject.

The secondary objective is to evaluate the tolerability and local and systemic effects of transdermal Human Insulin if any.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a serum protein HbA1c of less than 6.
2. The subject is willing and able to read, understand the Subject Information Sheet and provide written informed consent.
3. The subject has a body mass index (BMI) within 18-50 kg/m2.
4. The subject is in otherwise good health as determined by medical history and physical examination.
5. The subject is a non-smoker.
6. The subject must agree to continue with daily serum glucose testing by means of a wearable blood glucose for the pharmacokinetic assessments.
7. The subject is willing and able to comply with all testing and requirements defined in the protocol.
8. The subject is willing and able to return to the study site for all visits.

Exclusion Criteria:

1. The subject has any relevant deviations from normal other than blood glucose in physical examination, electrocardiogram (ECG), or clinical laboratory tests, as evaluated by the investigator.
2. The subject has had a clinically significant illness within 30 days preceding entry into this study.
3. The subject has a history of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease.
4. The subject has a known allergy or history of hypersensitivity to Human Insulin or similar modified Insulin compounds.
5. The subject has used any prescription medication that may interfere with the evaluation of study medication.
6. The subject has donated or lost a significant volume of blood (>450 mL) within four (4) weeks of the study, and their Haemoglobin concentration and haematocrit have not returned to within 5% of normal.
7. The subject has a history of substance abuse or a current positive urine drug screen or urine alcohol test.
8. Alcohol consumption greater than community norms (i.e. more than 21 standard drinks per week for males).
9. Subjects who have received an investigational drug or have used an investigational device in the 30 days prior to study entry

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 7 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William D. Kirsh, D.O., M.P.H., Principal Investigator — Langford Research Institute
Locations (1):
- Langford Research Institute, Palm Beach Gardens, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects ("Ss") were recruited by word-of-mouth and attended a study orientation where the study participation expectations were discussed and the informed consent forms provided. Ss underwent a health screening to ascertain healthy, non diabetic status.
Pre-assignment Details: 7 Volunteers were asked to undergo a physical exam including a complete metabolic panel via blood sample.
Groups:
- Main Experimental: 7 Subjects. Each subject received doses applied to the skin of 0.075 IUs / Kilogram Body Weight, 0.1 IUs/Kilogram Body Weight and 0.15 IUs /Kilogram Body Weight
  Human insulin: Human Insulin from recombinant source delivered in a solution capable of enabling transdermal delivery formulated at 100 IU/mL of delivery vehicle.
Period: Overall Study
Arm/Group | Main Experimental
Started | 7
Completed | 5
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Main Experimental
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Average Untreated Serum Glucose [Mean (Full Range); unit: mg/dL] | 96.4 [87 to 103]

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Serum Glucose in mg/dL as a Response to Small Doses (0.075 to 0.15 IUs/Kg) Human Insulin Averaged Per Subject
Description: An Average Postprandial serum glucose measured by the Continuous Glucose Monitor as a response to a single dose of Human Insulin averaged (Mean) for each Subject. Data is reported in mg/dL. The Average reported was a comparison from Baseline (Day 1) and up to 3.5 hours following each dose (assessed at Day 1 - Baseline, Day 2 - Dose 1, Day 3 - Dose 2, and Day 4 - Dose 3)"
Time Frame: Pre-dose Baseline & a Mean of readings over 3.5 hours
Population: We recruited and entered 7 healthy individuals into the study. We did not include data from 2 Subjects due to non-compliance with the protocol.
Measure: Mean (Full Range); unit: mg/dL
Groups:
- Dose 1: Each subject will receive doses applied to the skin of 0.075 IUs / Kilogram Body Weight,
  Human insulin: Human Insulin from recombinant source delivered in a solution capable of enabling transdermal delivery formulated at 100 IU/mL of delivery vehicle.
- Dose 2: Each subject will receive doses applied to the skin of 0.10 IUs / Kilogram Body Weight.
  Human insulin: Human Insulin from recombinant source delivered in a solution capable of enabling transdermal delivery formulated at 100 IU/mL of delivery vehicle.
- Dose 3: Each subject will receive doses applied to the skin of 0.15 IUs / Kilogram Body Weight.
  Human insulin: Human Insulin from recombinant source delivered in a solution capable of enabling transdermal delivery formulated at 100 IU/mL of delivery vehicle.
Arm/Group | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 5 | 5 | 5
mg/dL | 3.8 [-3 to 6] | -1.8 [-5 to 1] | 7 [-3 to 9]
Statistical Analysis 1: Comparison: Dose 1 vs Dose 2 vs Dose 3; Glucose was monitored by means of a wearable Continuous Glucose Monitor for several days prior to, during and post dosing. Measurements were gathered for each subject and averaged within-subject data. Our null hypothesis was that post prandial serum glucose would not vary significantly from their baseline values; Test type: Superiority; p = 0.000016, ANOVA; Degrees of Freedom = 5

2. Primary Outcome: Daily Average Serum Glucose Measured in mg/dL as a Response to Small Doses (0.075 to 0.15 IUs/Kg) Human Insulin
Description: Daily average serum glucose measured by the Continuous Glucose Monitor in measured in mg/dL as a response to a single dose of Human Insulin and reported by the Freestyle 14-day software. Data was collected 4 times an hour throughout the test period and across doses. The prandial segments were included in this average. Data is reported in mg/dL by subject.
Time Frame: 72 hours
Population: 7 healthy volunteers were recruited. Data from 2 of the subjects was not included, in both cases because of lack of compliance with device polling instructions. Subjects were directed to poll the sensor at least every 8 hours and follow a typical 3 meal schedule and these 2 subjects were unable to comply and or had device issues.
Measure: Mean (Full Range); unit: mg/dL Serum Glucose
Groups:
- Subject 1; Subject 2; Subject 4; Subject 5; Subject 6: Subject received doses applied to the skin of 0.075, 0.10 and 0.15 IUs / Kilogram Body Weight per dose.
  Human insulin: Human Insulin from recombinant source delivered in a solution capable of enabling transdermal delivery formulated at 50 IU/mL of delivery vehicle.
Arm/Group | Subject 1 | Subject 2 | Subject 4 | Subject 5 | Subject 6
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
mg/dL Serum Glucose | 95 [94 to 95] | 99 [98 to 101] | 85 [85 to 85] | 89 [87 to 93] | 103 [101 to 105]
Statistical Analysis 1: Comparison: Subject 1 vs Subject 2 vs Subject 4 vs Subject 5 vs Subject 6; Subject received doses applied to the skin of 0.075, 0.10 and 0.15 IUs / Kilogram on successive days. The Subject's average Serum Glucose for these 3 days were compared against the Subject's baseline unmedicated Serum Glucose on non-dosed days; Test type: Superiority; p = 0, t-test, 1 sided; Degrees of Freedom = 3
Statistical Analysis 2: Comparison: Subject 2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.000003, t-test, 1 sided
Statistical Analysis 3: Comparison: Subject 4; Test type: Superiority; p = 0.000002, t-test, 1 sided; Degrees of Freedom = 3
Statistical Analysis 4: Comparison: Subject 5; Test type: Superiority; p = 0.000035, t-test, 1 sided; Degrees of Freedom = 3
Statistical Analysis 5: Comparison: Subject 6; Test type: Superiority; p = 0.000004, t-test, 1 sided; Degrees of Freedom = 3

3. Secondary Outcome: OECD Acute Dermal Irritation/Corrosion Score According to to the Organisation for Economic Co-operation and Development (OECD) Guideline for Testing of Chemicals No. 404
Description: The skin at the application site will be assessed at each Clinic Visit by the investigator and/or Study Nurse. Any dermal irritation will be scored according to to the Organisation for Economic Co-operation and Development (OECD) Guideline for Testing of Chemicals No. 404, adopted 17th July, 1992: "Acute Dermal Irritation/Corrosion" and any score of 0 or greater will be reported.
  The Guideline is a scale of from Zero (No erythema or edema), 1: Very slight, 2: Well-defined erythema/Slight edema (edges of area well-defined by definite raising), 3: Moderate to severe erythema/Moderate edema (raised approximately 1 mm) to 4: Severe erythema (beet redness) to eschar formation preventing grading / Severe edema (raised more than 1 mm, extending beyond area of exposure). The higher the score the worse the erythema or edema, so a score of 0 is very good and a score of 4 is very bad.
Time Frame: 20 Days
Measure: Median (Full Range); unit: units on a scale
Groups:
- Main Experimental: Each subject will receive doses applied to the skin of 0.075 IUs / Kilogram Body Weight, 0.1 IUs/Kilogram Body Weight and 0.15 IUs /Kilogram Body Weight
  Human insulin: Human Insulin from recombinant source delivered in a solution capable of enabling transdermal delivery formulated at 100 IU/mL of delivery vehicle.
  Any subject scored as 1 or higher on the OECD Acute Dermal Irritation/Corrosion Scale will be counted.
Arm/Group | Main Experimental
Number analyzed (Participants) | 5
units on a scale | 0 [0 to 0]
Statistical Analysis 1: Comparison: Main Experimental; Test type: Superiority; p = 0, ANOVA

ADVERSE EVENTS:
Time Frame: 21 Days
Arm/Group | Main Experimental
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT04857320/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT04857320/SAP_001.pdf